CLINICAL TRIAL: NCT06448169
Title: Observational Study on the Sensitivity of Neoadjuvant Immunotherapy in Early Triple-Negative Breast Cancer Based on High-Resolution Dynamic Immune Signature Analysis
Brief Title: Observational Study on the Sensitivity of Neoadjuvant Immunotherapy in Early Triple-Negative Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Zhi Gang, M.D., Shandong University
Other Study IDs: STNBC001
Record Dates: First submitted 2024-05-12; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Triple Negative Breast Cancer; Neoadjuvant Immunotherapy; Sensitivity
Keywords: Sensitivity; Neoadjuvant Immunotherapy; Triple-Negative Breast Cancer; Dynamic Immune Signature Analysis
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Hypersensitivity | interventions — Immune Checkpoint Inhibitors; tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Utilize deep sequencing technology to capture the molecular characteristics of the TCR immunome pool in the peripheral blood of patients with triple-negative breast cancer at different time points before and after neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 inhibitor combined with neoadjuvant chemotherapy
  Other Names: Tislelizumab

SUMMARY:
Studies have reported that tumors with the same immunogenic mutations may induce T cell receptor (TCR) domains with similar antigen recognition functions. By assembling the complementarity-determining region 3 (CDR3) of TCRs from RNA-seq data and correlating them with 9142 samples from TCGA data, an in-depth analysis of the TCR pool in the tumor microenvironment found a strong correlation between the CDR3 sequences of tumor-infiltrating T cells and tumor mutation burden. Fairfax et al. found that in patients responding to tumor immunotherapy, the TCR immune pool of CD8+ T cells produces many clones with extremely high abundance (exceeding 0.5%) . Cader et al. also found significant changes in the TCR immune pool of patients with Hodgkin's lymphoma responding to PD-1 tumor immunotherapy. Based on these theoretical foundations, evaluating the dynamic changes of the TCR immune pool is expected to be used to analyze the immune characteristics and changes in diseases such as malignant tumors.

DETAILED DESCRIPTION:
I. Background, Approximately 12-17% of breast cancer patients suffer from triple-negative breast cancer (TNBC) , which is prone to visceral and central nervous system metastases, poses significant therapeutic challenges, and has poor prognosis. Clinically starting with early TNBC, strengthening precise and individualized treatment, and reducing the risk of recurrence and metastasis are effective methods to improve the survival rate of TNBC patients.

The optimization of neoadjuvant therapy regimens has always been a research hotspot. Traditional neoadjuvant therapy regimens are primarily based on chemotherapy. The KEYNOTE-522 study showed that traditional chemotherapy combined with PD-1 inhibitors could significantly increase the pCR (pathological complete remission) rate, improving by 13.6% (64.8% vs 51.2%, P=0.00055) and reducing the risk of recurrence. However, this treatment also brings inevitable immune-related adverse events (AEs), with an overall AE incidence rate of 43.6%, a 3-5 grade AE incidence rate of 14.9%, and a fatal AE rate of 0.3%. Many immune-related AEs are lifelong, such as hypothyroidism. Therefore, how to precisely select immunologically sensitive patients for immunotherapy, while administering chemotherapy only to those who are immunologically insensitive, to avoid unnecessary immune-related AEs? How to predict patients who may experience severe immune-related adverse reactions early? These are urgent clinical issues that need to be addressed. Meanwhile, the mechanism of immunotherapy resistance remains unclear.

Studies have reported that tumors with the same immunogenic mutations may induce T cell receptor (TCR) domains with similar antigen recognition functions. By assembling the complementarity-determining region 3 (CDR3) of TCRs from RNA-seq data and correlating them with 9142 samples from TCGA data, an in-depth analysis of the TCR pool in the tumor microenvironment found a strong correlation between the CDR3 sequences of tumor-infiltrating T cells and tumor mutation burden. Fairfax et al. found that in patients responding to tumor immunotherapy, the TCR immune pool of CD8+ T cells produces many clones with extremely high abundance (exceeding 0.5%). Cader et al. also found significant changes in the TCR immune pool of patients with Hodgkin's lymphoma responding to PD-1 tumor immunotherapy. Based on these theoretical foundations, evaluating the dynamic changes of the TCR immune pool is expected to be used to analyze the immune characteristics and changes in diseases such as malignant tumors.

Research Aim and Significance This study aims to utilize deep sequencing technology to capture the molecular characteristics of the TCR immunome pool in the peripheral blood of patients with triple-negative breast cancer at different time points before and after neoadjuvant therapy. By combining artificial intelligence analysis algorithms, the investigators aim to accurately screen the patient population that will benefit from neoadjuvant immunotherapy for triple-negative breast cancer, avoid the occurrence of severe immune-related AEs, and explore the mechanisms of resistance to immunotherapy, ultimately achieving individualized and precise immunotherapy.

Research Content Analyze the changing characteristics of the TCR dynamic molecular group before neoadjuvant therapy in patients with triple-negative breast cancer, and compare the benefited and non-benefited patients receiving neoadjuvant therapy to screen for the population that will benefit from neoadjuvant immunotherapy for triple-negative breast cancer.

Analyze the changing characteristics of the TCR dynamic molecular population during neoadjuvant therapy in patients with triple-negative breast cancer, and compare patients who experience severe immune-related adverse events with those who do not, in order to prevent and detect severe immune-related adverse events early.

Analyze the changing characteristics of the TCR dynamic molecular population in patients with neoadjuvant therapy resistance for triple-negative breast cancer, examine the immune characteristics of resistant patients, and explore the mechanisms of resistance to immunotherapy.

Research Design

1. Randomized Control Method: This is a non-randomized controlled, single-arm, open-label design.
2. Sample Size: This study plans to enroll 200 participants.
3. Study Population: Early-stage triple-negative breast cancer patients receiving neoadjuvant therapy with PD-1 inhibitors combined with chemotherapy.
4. Treatment Factors (Placebo, Drugs, or Other Interventions): Neoadjuvant therapy drugs include PD-1 inhibitors (200mg, intravenous infusion, administered on day 1 of each cycle, with 21 days as a cycle), albumin-bound paclitaxel (260 mg/m2, intravenous infusion, administered on day 1 of each cycle, with 21 days as a cycle), and carboplatin (AUC 4, administered on day 1 of each cycle, with 21 days as a cycle).
5. Primary/Secondary Observation Indicators: Pathological complete response rate, clinical response rate, immune-related adverse events, and drug resistance.
6. Safety and Effectiveness Evaluation Indicators: Perform imaging examinations every 2 cycles during the treatment period to evaluate efficacy, based on the RECIST 1.1 standard. After completing 6 cycles of neoadjuvant therapy, surgery will be performed, and pathological evaluation of the therapeutic effect will be conducted.

Inclusion/Exclusion Criteria and Withdrawal/Termination Criteria of the Subjects

1. Recognized Diagnostic Criteria for the Target Disease: Pathological examination by core needle biopsy.
2. Inclusion Criteria:

1) Age: 18-60 years old; 2) Histologically confirmed triple-negative breast cancer, with immunohistochemistry showing ER <1%, PR <1%, HER2-negative (IHC 0 or 1+; or IHC 2+ ISH-negative); 3) Imaging-confirmed non-metastatic disease; 4) Clinical efficacy can be evaluated according to RECIST criteria; 5) European Functional Handicap Scale (MRC) of 0-2; 6) The investigator determines that the treatment is tolerable based on the patient's organ function level; 7) Volunteers willing to participate in this study, sign the informed consent, have good compliance, and are willing to cooperate with follow-up.

3. Exclusion Criteria:

1. Immunohistochemistry showing HER2-positive (IHC 3 or IHC 2 ISH-amplified);
2. Previously treated;
3. Severe dysfunction of important organs such as heart, liver, and kidneys;
4. Patients with diseases unsuitable for immunotherapy;
5. Known allergy history to any component of the drugs in this regimen;
6. History of immune deficiency, including HIV-positive, HCV, active hepatitis B, or other acquired or congenital immune deficiency diseases, or a history of organ transplantation;
7. Any cardiac disease, including: ① Medically treated or clinically significant arrhythmias; ② Myocardial infarction; ③ Heart failure; ④ Any other cardiac disease judged by the investigator as unsuitable for participation in this trial;
8. Pregnant or lactating women, fertile women with positive baseline pregnancy test or those unwilling to take effective contraceptive measures during the entire trial;
9. According to the investigator's judgment, there are accompanying diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension uncontrollable by drugs, severe diabetes, active infections, etc.);
10. Long-term use of drugs that affect the components of peripheral blood immune cells, such as recombinant human erythropoietin, recombinant human granulocyte colony-stimulating factor, recombinant human interleukin, or Likejun tablets;
11. Received immunosuppressive therapy within 2 weeks;
12. Hematological precancerous diseases, such as myelodysplastic syndrome, and coagulation disorders.

4. Have high-risk populations been excluded? Yes; 5. Have interfering factors been excluded? Yes; 6. Withdrawal/Termination Criteria:

1. The subject withdraws the informed consent and requests withdrawal;
2. Medical imaging or clinical progression;
3. Any clinical adverse event, abnormal laboratory test, or other medical condition occurs, leading to the possibility that continued medication may no longer benefit the subject;
4. Serious violation of the trial protocol, and the investigator assesses that treatment should be terminated;
5. Pregnancy occurs during the study;
6. Other reasons why the investigator believes that drug treatment cannot be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old;
2. Histologically confirmed triple-negative breast cancer, with immunohistochemistry showing ER <1%, PR <1%, HER2-negative (IHC 0 or 1+; or IHC 2+ ISH-negative);
3. Imaging-confirmed non-metastatic disease;
4. Clinical efficacy can be evaluated according to RECIST criteria;
5. European Functional Handicap Scale (MRC) of 0-2;
6. The investigator determines that the treatment is tolerable based on the patient's organ function level;
7. Volunteers willing to participate in this study, sign the informed consent, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Immunohistochemistry showing HER2-positive (IHC 3 or IHC 2 ISH-amplified);
2. Previously treated;
3. Severe dysfunction of important organs such as heart, liver, and kidneys;
4. Patients with diseases unsuitable for immunotherapy;
5. Known allergy history to any component of the drugs in this regimen;
6. History of immune deficiency, including HIV-positive, HCV, active hepatitis B, or other acquired or congenital immune deficiency diseases, or a history of organ transplantation;
7. Any cardiac disease, including: ① Medically treated or clinically significant arrhythmias; ② Myocardial infarction; ③ Heart failure; ④ Any other cardiac disease judged by the investigator as unsuitable for participation in this trial;
8. Pregnant or lactating women, fertile women with positive baseline pregnancy test or those unwilling to take effective contraceptive measures during the entire trial;
9. According to the investigator's judgment, there are accompanying diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension uncontrollable by drugs, severe diabetes, active infections, etc.);
10. Long-term use of drugs that affect the components of peripheral blood immune cells, such as recombinant human erythropoietin, recombinant human granulocyte colony-stimulating factor, recombinant human interleukin, or Likejun tablets;
11. Received immunosuppressive therapy within 2 weeks;
12. Hematological precancerous diseases, such as myelodysplastic syndrome, and coagulation disorders.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: early stage triple negative breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | after operation, an average of 5 months
  patients with pCR/all patients *100%

SECONDARY OUTCOMES:
clinical response rate | before operation,an average of 5 months
  patients with cCR/all patients *100%
immune-related adverse events | during treatment, ,an average of 5 months
  AE related to immune therapy
drug resistance | during treatment,,an average of 5 months
  immune therapy resistance, tumor no reaction to immunotherapy

IPD SHARING:
Plan to Share IPD: Undecided